CLINICAL TRIAL: NCT00073814
Title: An Efficacy, Safety, and Tolerability Study of Daily Dosing With Levalbuterol, Racemic Albuterol, and Placebo in Pediatric Subjects With Asthma
Brief Title: Study of Daily Dosing With Levalbuterol, Racemic Albuterol, and Placebo in Pediatric Subjects With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 051-354
Record Dates: First submitted 2003-12-09; First posted 2003-12-10 (Estimated); Last update posted 2012-02-22 (Estimated); Status verified 2012-02

CONDITIONS: Asthma
Keywords: levalbuterol; pediatric; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): levalbuterol MDI 90 mcg QID
  Interventions: Drug: Levalbuterol tartrate MDI
- 2 (Active Comparator): racemic albuterol MDI 190 mcg QID
  Interventions: Drug: racemic albuterol MDI
- 3 (Placebo Comparator): Placebo MDI QID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levalbuterol tartrate MDI — levalbuterol MDI 90 mcg QID
  Other Names: Xopenex MDI
  Arms: 1
Drug: racemic albuterol MDI — racemic albuterol MDI 180 mcg QID
  Arms: 2
Drug: Placebo — Placebo MDI QID
  Arms: 3

SUMMARY:
Study of Daily Dosing with Levalbuterol, Racemic Albuterol, and Placebo in Pediatric Subjects with Asthma

DETAILED DESCRIPTION:
This was a Phase III, double-blind, randomized, placebo- and active-controlled, multicenter, parallel-group study of up to 6 weeks in duration. Seven days of QID single-blind, placebo administration (via HFA MDI) was followed by 28 days of QID, double-blind treatment. A follow-up visit was required only for subjects who had, in the opinion of the investigator, a clinically significant finding at Visit 6 /ET that would put the subject at risk. A final follow up phone evaluation was conducted 7 days after the completion of Visit 6/ET. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria

* Subject and subject's p/l guardian must be willing and able to comply with the study procedures and visit schedules
* Subject, male or female, between the ages of 4 to 11 yrs
* Female subjects 8 yrs or older will have a negative serum pregnancy test
* Must have a documented diagnosis of asthma for a minimum of 6 months prior to study start
* Must have stable baseline asthma and have been using a B-adrenergic agonist, and/or anti-asthma anti-inflammatory medication, and/or over-the-counter asthma medication for at least 6 mos. prior to study start
* Must be in good health with the exception of reversible airways disease and not suffering from any chronic condition that might affect their respiratory function
* Must have a chest X-ray that is not diagnostic of pneumonia, atelectasis, pulmonary fibrotic disease, pneumothorax, chronic obstructive pulmonary disease etc
* Subject's p/l guardian must be able to complete the diary cards and medical event calendars reliably on a daily basis, understand dosing instructions and questionnaire completion, and demonstrate how to use the MiniWright PEF meter

Exclusion Criteria

* Female subject who is pregnant or lactating
* Have participated in an investigational drug study within 30 days prior to study start, or who is currently participating in another clinical trial
* Schedule prevents him or her from taking the first daily dose of study medication and/or starting study visits before 9 AM
* Have travel commitments during the study that would interfere with trial measurements or compliance or both
* Have a history of hospitalization for asthma within 60 days prior to study start, or who is scheduled for in-patient hospitalization, including elective surgery during the course of the trial
* Have a known sensitivity to levalbuterol or racemic albuterol, or any of the excipients contained in any of these formulations
* Subject using any prescription drug with which albuterol sulfate administration is contraindicated
* Have currently diagnosed life-threatening asthma defined as a history of asthma episodes requiring intubation, associated with hypercapnia, respiratory arrest, or hypoxic seizures within 3 mos. prior to study start
* Have a history of cancer
* Subject with hyperthyroidism, diabetes, hypertension, cardiac diseases or seizure disorders that currently are not well controlled by medication or that may interfere with the successful completion of this protocol
* Have a history of substance abuse or drug abuse within 12 months preceding V1 or a positive urine drug screening at study start
* Have a documented history of bronchopulmonary aspergillosis or any form of allergic alveolitis
* Has suffered from a clinically significant upper or lower respiratory tract infection in the 2 wks prior to study start
* Have a history of cigarette smoking or use of any tobacco products
* Subject who is a relative of a staff member

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2002-12; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
was peak percent change in FEV1 from visit predose averaged over the double-blind period | Week 0, 2, 4

SECONDARY OUTCOMES:
under the FEV1 percent change from visit predose curve averaged over the double-blind period | Week 0, 2, 4
peak change and peak percent change in FEV1 from visit predose to each visit | Week 0, 2, 4
peak change in FEV1 from visit predose to each visit | Week 0, 2, 4
peak percent change in FEV1 from study baseline over the double blind period | Week 0, 2, 4
time to peak change | Week 0, 2, 4
peak percent of predicted FEV1 at each visit and over the double-blind period | Week 0, 2, 4
area under the FEV1 percent change from predose curve at each visit | Week 0, 2, 4
area under the FEV1 percent change from study baseline curve at each visit and averaged over the double-blind period | Week 0, 2, 4
percent of predicted FEV1 AUC at each visit | Week 0, 2, 4
percent change in predose FEV1 from study baseline at each visit | Week 0, 2, 4
number and percent of responders | Week 0, 2, 4
time to onset of response and duration of response | Week 0, 2, 4

CONTACTS AND LOCATIONS:
Locations (45):
- United States (45):
  - Adolescent & Pediatric Associates, PC, Montgomery, Alabama
  - The Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - Integrated Research Group, Corona, California
  - Allergy & Asthma Specialists Medical Group, Huntington Beach, California
  - Asthma, Allergy & Respiratory Care Center, Long Beach, California
  - Madera Family Medical Group, Madera, California
  - Southern California Research, Mission Viejo, California
  - CHOC, PSF, AMC Disision of Allergy, Asthma & Immunology, Orange, California
  - Clinical Trials of Orange County, Orange, California
  - Allergy Associates Medical Group, San Diego, California
  - West Coast Clinical Trials, Inc., Signal Hill, California
  - Allergy & Asthma Medical Group of Diablo Valley, Inc., Walnut Creek, California
  - Asthma & Allergy Associates, Colorado Springs, Colorado
  - National Jewish Medical & Research Center, Denver, Colorado
  - The Allergy & Asthma Clinical Research Center, Lawrenceville, Georgia
  - Aeroallergy Research Laboratories of Savannah, Inc., Savannah, Georgia
  - Department of Pediatric Critical Care, Kosair Children's Hospital, Louisville, Kentucky
  - The Pediatric Clinic, Bogalusa, Louisiana
  - Doctor's Care, New Orleans, Louisiana
  - Dolby Providers, Inc, New Orleans, Louisiana
  - Radiant Research, Bridgeton, Missouri
  - Essex-Morris Pediatric Group, Livingston, New Jersey
  - Princeton Center for Clinical Research, Princeton, New Jersey
  - Summit Pediatric Pulmonology, Summit, New Jersey
  - University of New Mexico, Health Sciences Center, Albuquerque, New Mexico
  - Pulmonary Associates of Mobile, PC, Ithaca, New York
  - Regional Allergy & Asthma Consultants, PA, Asheville, North Carolina
  - Pediatric Associates of Mt. Carmel, Cincinnati, Ohio
  - University Hospitals of Cleveland, Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Dr. Senders & Associates, University Heights, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Allergy & Asthma and Dermatology Research Center, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Bellevue Pediatric Association, Pittsburgh, Pennsylvania
  - Allergy & Asthma Consultants, Mt. Pleasant, South Carolina
  - Allergy, Asthma & Sinus Center, PC, Knoxville, Tennessee
  - Vanderbilt University ASAP Research, Nashville, Tennessee
  - Pediatric Allergy/Immunology Associates, Dallas, Texas
  - North Texas Institute for Clinical Trials, Fort Worth, Texas
  - Allergy & Asthma Associates, Houston, Texas
  - Breath of Life Research Institute, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - PI- Coor Clinical Research, LLC, Burke, Virginia
  - Allergy & Asthma Associates, Kirkland, Washington